CLINICAL TRIAL: NCT03418220
Title: Comparison of Cytokine Profiles in Aqueous Humor of Patients With Age Related Macular Degeneration (AMD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 69HCL17_0544; 2017-A02365-48 (Other: ANSM)
Record Dates: First submitted 2018-01-25; First posted 2018-02-01 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Macular Degeneration, Age-Related
Keywords: Age related Macular Degeneration; Atrophy; Inflammation; Cytokines; test LUMINEX®
MeSH Terms: conditions — Macular Degeneration; Atrophy; Inflammation | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- AMD early / intermediate (Other): A blood and aqueous humor sample will be taken during cataract surgery in patients with AMD early / intermediate
  Interventions: Other: blood and aqueous humor sampling
- AMD exudative (Other): A blood and aqueous humor sample will be taken during cataract surgery in patients with AMD exudative
  Interventions: Other: blood and aqueous humor sampling
- AMD atrophic (Other): A blood and aqueous humor sample will be taken during cataract surgery in patients with AMD atrophic
  Interventions: Other: blood and aqueous humor sampling
- control group (Other): A blood and aqueous humor sample will be taken during cataract surgery in patients with cataract (control group)
  Interventions: Other: blood and aqueous humor sampling

INTERVENTIONS:
Other: blood and aqueous humor sampling — The blood sample will be centrifuged. The plasma will be recovered. Plasma and aqueous humor will be frozen and stored at -80° Celsius. The search of 27 markers of inflammation will be performed by the kit LUMINEX Bio-rad (Bio-Rad, M500KCAF0Y).

SUMMARY:
Age-related macular degeneration (AMD) affects 2 million people in France. It characterized by progressive degeneration of the central area of the retina allowing detailed vision. It is the main cause of irreversible blindness in France. All patients initially present an early form, the latter can evolve in two different ways: the atrophic form, which progresses slowly, and the exudative or neovascular form, of more rapid evolution. While the treatment of exudative AMD has improved dramatically in recent years, there is currently no therapy for atrophic AMD. Recently, it has been demonstrated in atrophic AMD, an accumulation of inflammatory cells, macrophages, in the sub-retinal space. This space is located between the pigment epithelium (PE) and the photoreceptors. It is physiologically devoid of immune cells (immune privilege). Macrophages will secrete many pro-inflammatory molecules, such as cytokines. It has been shown in mouse models that some cytokines (IL-1beta, IL6 et TNFalpha) have a deleterious role on (PE) and photoreceptors. The identification of specific cytokines in the aqueous humor of patients with atrophic AMD would help to better understand this disease and consider potential targeted therapies. This study will be conducted in the ophthalmology department of the Croix-Rousse Hospital in Lyon. 80 patients will be recruited and divided into 4 groups: three experimental groups of 20 patients with : Early / Intermediate AMD, atrophic AMD or exudative AMD, and one control group of 20 patients without signs of AMD. Assays of the markers will be performed using the Luminex® technique on aqueous humor and blood samples collected for all patients during cataract surgery. The concentrations obtained in the aqueous humor will be normalized on their respective blood levels in order to confirm the intraocular secretion of these markers,. The identification of particular cytokine profiles in atrophic AMD compared to other forms of AMD would support emerging hypotheses of involvement of specific inflammatory cells in this pathology. There is currently no treatment available for atrophic AMD. If molecular screening identifies one or more specific biomarkers, targeted therapy may be considered.

ELIGIBILITY:
Inclusion Criteria:

* • GENERAL CRITERIA
* Man or woman with age over 60 years,
* Informed, written and signed consent by the patient and the investigator (no later than the day of inclusion) and before any investigation required by the research,
* Patient affiliated with social security,
* Patient willing and able to return to all clinical visits to the study and complete all related procedures.

  • SPECIFIC CRITERIA
* Patient who need a cataract surgery,
* Patient presenting in both eyes:

the same type of AMD defined according to the international AREDS study modified (Ferris et al., 2013) no other ophthalmological pathology (control group).

Exclusion Criteria:

* • GENERAL CRITERIA
* Major patient under tutorship or curatorship or unable to express consent,
* Person deprived of liberty,
* Patient participating in an ongoing clinical trial during the inclusion visit,

  • SPECIFIC CRITERIA
* Patient with chronic ophthalmic pathologies other than cataract and AMD defined in the modified international AREDS study included in the eye (Ferris et al., 2013),
* Patient who participated in a clinical trial of an experimental drug for atrophic AMD,
* Patient taking systemically drugs with immunomodulatory action: immunosuppressants, immunomodulators, chemotherapy or corticosteroids,
* Patient with systemic diseases modifying his immune status,
* Patient with a history of diabetes,
* Patient who received an anti-inflammatory eye treatment in both eyes in the 6 months preceding the surgery,
* Patient having dynamic phototherapy on the included eye.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2017-11-22 (Actual); Primary Completion 2020-09-08 (Actual); Study Completion 2020-09-08 (Actual)

PRIMARY OUTCOMES:
Comparison of concentrations of intraocular inflammation markers between the group of patients with atrophic AMD and the control group. | day of surgery
  Aqueous humor sample will be collected during the cataract surgery in patient with atrophic AMD and in patient of control group. In order to identify and quantify intraocular inflammation markers in samples, LUMINEX® Multiplex analysis of the samples will be done by the Bio-Plex Pro Human Cytokine 27-Plex Panel (Bio-Rad, M500KCAF0Y). This test allow identification of one or more of the following 27 inflammation markers: basic FGF, Eotaxin, G-CSF, GM-CSF, interferon (IFNγ), interleukin (IL1β, IL1ra, IL2, IL4, IL5, IL6, IL7, IL8, IL9, IL10, IL12, IL13 , IL15, IL17), IP10, MCP1, MIP1α, MIP1β, PDGF-BB, RANTES, TNFα and Vascular Endothelial Growth Factor (VEGF).

SECONDARY OUTCOMES:
Comparison of the concentration ratios of inflammation marker [aqueous humor / blood] between the group of patients with atrophic AMD and the control group. | day of surgery
  Aqueous humor sample and the blood sample will be collected during the cataract surgery in patient with atrophic AMD and in patient of control group. In order to identify and quantify inflammation markers, LUMINEX® Multiplex analysis of the samples will be done by the Bio-Plex Pro Human Cytokine 27-Plex Panel (Bio-Rad, M500KCAF0Y).
  For each identified intraocular inflammatory marker, the ratio between the level of expression in the aqueous humor sample and the level of expression in the blood sample will be calculated.
  Each ratio will be compared between patients with atrophic AMD and patients of control group.
Comparison of the concentration ratios of inflammation marker [aqueous humor / blood] between the different stages of AMD: early / intermediate, exudative or atrophic | day of surgery
  Aqueous humor sample and the blood sample will be collected during the cataract surgery in patient with different stage of AMD : early / intermediate, exudative or atrophic.
  In order to identify and quantify inflammation markers, LUMINEX® Multiplex analysis of the samples will be done by the Bio-Plex Pro Human Cytokine 27-Plex Panel (Bio-Rad, M500KCAF0Y). For each identified intraocular inflammatory marker, the ratio between the level of expression in the aqueous humor sample and the level of expression in the blood sample will be calculated and compared between different stages of AMD: early / intermediate, exudative or atrophic.
Comparison of the concentration ratios of inflammation marker [aqueous humor / blood] between the different types of atrophic AMD defined by autofluorescence exam (non-hyperautofluorescent or hyperautofluorescent form) | day of surgery
  Autofluorescence exam allows in vivo mapping of lipofuscin distribution. Lipofuscin is a fluorophore of the retinal pigment epithelium. Autofluorescence represents in gray scale the spatial distribution of lipofuscin, and reflect the metabolic activity of the retinal pigment epithelium. Autofluorescence exam allows classification in different types of atrophic AMD. Autofluorescence exam was performed for all patients at the first visit. Aqueous humor sample and blood sample will be collected during the cataract surgery. In order to identify and quantify inflammation markers, LUMINEX® Multiplex analysis of the samples will be done by the Bio-Plex Pro Human Cytokine 27-Plex Panel (Bio-Rad, M500KCAF0Y). For each identified intraocular inflammatory marker, the ratio between the level of expression in the aqueous humor sample and the level of expression in the blood sample will be calculated, and compared between the different types of atrophic AMD.
Comparison of the concentration ratios of inflammation marker [aqueous humor / blood] according to the macular atrophy area measured by autofluorescence in atrophic AMD. | day of surgery
  Macular atrophy area is measured at first visit in autofluorescent exam. Aqueous humor sample and the blood sample will be collected during the cataract surgery. In order to identify and quantify inflammation markers, LUMINEX® Multiplex analysis of the samples will be done by the Bio-Plex Pro Human Cytokine 27-Plex Panel (Bio-Rad, M500KCAF0Y). For each identified intraocular inflammatory marker, the ratio between the level of expression in the aqueous humor sample and the level of expression in the blood sample will be calculated, and compared between the different size of macular atrophy area.
Comparison of the concentration ratios of inflammation marker [aqueous humor / blood] according to the central retinal thickness measured by Optical Coherence Tomography (OCT) in atrophic AMD | day of surgery
  OCT define precisely the retinal structures and their locations. Aqueous humor sample and the blood sample will be collected during the cataract surgery. In order to identify and quantify inflammation markers, LUMINEX® Multiplex analysis of the samples will be done by the Bio-Plex Pro Human Cytokine 27-Plex Panel (Bio-Rad, M500KCAF0Y). For each identified intraocular inflammatory marker, the ratio between the level of expression in the aqueous humor sample and the level of expression in the blood sample will be calculated, and compared between the different thickness of retina measured by OCT .
Comparison of the concentration ratios of inflammation marker [aqueous humor / blood] according to the recognized risk factors of AMD | day of surgery
  ratios of [aqueous humor / blood] concentrations of inflammation markers will be compared on age, female sex, smoking (number of pack-years), obesity (body mass index)

CONTACTS AND LOCATIONS:
Overall Officials: Thibaud Mathis, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hôpital de la Croix-Rousse, Lyon, France

REFERENCES:
- [Background] Roubeix C, Nous C, Augustin S, Ronning KE, Mathis T, Blond F, Lagouge-Roussey P, Crespo-Garcia S, Sullivan PM, Gautier EL, Reichhart N, Sahel JA, Burns ME, Paques M, Sorensen TL, Strauss O, Guillonneau X, Delarasse C, Sennlaub F. Splenic monocytes drive pathogenic subretinal inflammation in age-related macular degeneration. J Neuroinflammation. 2024 Jan 17;21(1):22. doi: 10.1186/s12974-024-03011-z. PMID 38233865